CLINICAL TRIAL: NCT05303675
Title: The Effect of Education, Lymphedema Risk Scoring, and Progressive Upper Extremity Exercises on Strengthening the Self-care Skills of Women Who Have Breast Cancer Surgery
Brief Title: The Effect of Arm Exercises on Arm Oedema After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulseren MARAS (Other)
Responsible Party: Sponsor-Investigator, Gulseren MARAS, Research Assistant, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 710/2021
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female; Breast Cancer Lymphedema
Keywords: breast cancer; lymphedema; risk scoring; exercise; self-care
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Preoperative: An introductory information form will be filled out, and a lymphedema self-care and exercise booklet will be given.
  Postoperative: Patients will be applied Progressive Upper Limb Exercises and Muscle Relaxation Training (PULE-MRT), lymphedema upper extremity circumference measurement, and symptom alert model until discharge, and Muscle Relaxation Training will continue until discharge.
  Post-Discharge: They will be asked to record a diary at home. PULE-MRT will continue until day 15. The 15-day exercise program will continue for up to 3 months. Follow-up will be made by telephone according to the symptom alert model at the 1st, 2nd, and 3rd months, and at the end of the 3rd month, the breast cancer-related lymphedema self-care scale will be administered.
  Interventions: Other: exercise and training
- Control Group (No Intervention): Preoperative: Introductory information form will be filled out. Postoperative: Standard nursing care will be applied to the patients, lymphedema upper extremity circumference measurement and symptom alert model follow-up form will be applied.
  Post-Discharge: Lymphedema upper extremity circumference measurement will be explained to the patients before discharge, and they will be asked to record the 1st, 2nd, and 3rd months at home. Patients will be followed up by telephone according to the symptom alert model at the 1st, 2nd, and 3rd months, and at the end of the 3rd month, the breast cancer-related lymphedema self-care scale will be administered.

INTERVENTIONS:
Other: exercise and training — Preoperative: An introductory information form will be filled out, and a lymphedema self-care and exercise booklet will be given.
  Postoperative: Patients will be applied Progressive Upper Limb Exercises and Muscle Relaxation Training (PULE-MRT), lymphedema upper extremity circumference measurement, and symptom alert model until discharge, and Muscle Relaxation Training will continue until discharge.
  Post-Discharge: They will be asked to record a diary at home. PULE-MRT will continue until day 15. The 15-day exercise program will continue for up to 3 months. Follow-up will be made by telephone according to the symptom alert model at the 1st, 2nd, and 3rd months, and at the end of the 3rd month, the breast cancer-related lymphedema self-care scale will be administered.
  Arms: Intervention Group

SUMMARY:
In order to prevent lymphedema after breast surgery, patients are advised to know the risk factors for lymphedema and to avoid situations that may cause lymphedema, to perform active and passive arm exercises, to evaluate the affected area for lymphedema, to perform self-care and this should be under the self-management of the patients. Investigators think that this study will have a positive effect on the literature since there are no studies on risk scoring, the combined use of training and exercises to strengthen self-care skills in preventing the development of breast cancer-associated lymphedema. From this point of view, the study was planned as a randomized controlled experiment to examine the effects of preoperative lymphedema scoring and postoperative progressive upper extremity exercises on upper extremity function and self-care in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female gender,
* Between 18-65 years old
* BMI ≤30 kg/m2
* Axillary lymph node dissection (removal of at least 2 lymph nodes),
* No history of cancer other than breast cancer,
* Does not have any chronic disease (such as diabetes mellitus, hypertension, chronic obstructive pulmonary disease) that prevents exercise
* No previous diagnosis of lymphedema,
* Not pregnant or breastfeeding during the study,
* Individuals who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Total (simple) mastectomy,
* History of bilateral lymph node dissection,
* Lymphedema (difference >2 cm with an intact extremity)
* Individuals who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female gender, breast cancer surgery
Enrollment: 40 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
arm circumference measurement | 1st month
  Change from baseline in arm circumference at 1 month. Arm circumference measurement:An increase of 1 cm or more in the circumference of the affected arm compared to the healthy side and an increase of 2 cm or more for late detection of lymphedema indicates the presence of lymphedema.
arm circumference measurement | 2nd month
  Change from baseline in arm circumference at 2 month. Arm circumference measurement: An increase of 1 cm or more in the circumference of the affected arm compared to the healthy side and an increase of 2 cm or more for late detection of lymphedema indicates the presence of lymphedema.
arm circumference measurement | 3nd month
  Change from baseline in arm circumference at 3 month. Arm circumference measurement: An increase of 1 cm or more in the circumference of the affected arm compared to the healthy side and an increase of 2 cm or more for late detection of lymphedema indicates the presence of lymphedema.
lymphedema symptom | 1rd month
  Change from baseline in the number of lymphedema symptoms according to the 'Symptom Warning Model For Lymphedema' at 1-month. 'Symptom Warning Model For Lymphedema':The model consists of 17 symptoms and Yes/No response components. Patients with less than 15% of 17 symptoms are defined as low risk, 15-49% at medium risk, and patients with more than 50% symptoms are defined as high risk.
lymphedema symptom | 2rd month
  Change from baseline in the number of lymphedema symptoms according to the 'Symptom Warning Model For Lymphedema' at 2-month. 'Symptom Warning Model For Lymphedema':The model consists of 17 symptoms and Yes/No response components. Patients with less than 15% of 17 symptoms are defined as low risk, 15-49% at medium risk, and patients with more than 50% symptoms are defined as high risk.
lymphedema symptom | 3rd month
  Change from baseline in the number of lymphedema symptoms according to the 'Symptom Warning Model For Lymphedema' at 3-month. 'Symptom Warning Model For Lymphedema':The model consists of 17 symptoms and Yes/No response components. Patients with less than 15% of 17 symptoms are defined as low risk, 15-49% at medium risk, and patients with more than 50% symptoms are defined as high risk.
self-care | 3rd month
  The number of participants with a high self-care score according to the 'Breast Cancer-Related Lymphedema Self-Care Scale'. 'Breast Cancer-Related Lymphedema Self-Care Scale': The lowest 31, the highest 124 points are taken from the scale. Higher scores indicate better self-care.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No